CLINICAL TRIAL: NCT03068130
Title: An Extended Access Program to Assess Long-term Safety of Bardoxolone Methyl in Patients With Pulmonary Hypertension
Brief Title: Extended Access Program to Assess Long-term Safety of Bardoxolone Methyl in Patients With Pulmonary Hypertension RANGER
Acronym: RANGER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The company determined that continued exposure of these high-risk PH patients to clinic or in-person visits during the COVID pandemic presented an unacceptable risk.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTA 402-C-1602
Record Dates: First submitted 2017-02-22; First posted 2017-03-01 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension; Pulmonary Hypertension; PH; PAH; Bardoxolone methyl; 6-minute walk distance; CDDO-ME; RTA 402; LARIAT; CATALYST; RANGER
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — bardoxolone methyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bardoxolone methyl 10 mg (Experimental): Bardoxolone methyl will be administered orally once daily at 10 mg until it becomes commercially available. Dose de-escalation (down to 5 mg) is permitted during the study, if indicated clinically.
  Interventions: Drug: Bardoxolone methyl

INTERVENTIONS:
Drug: Bardoxolone methyl — Capsules of Bardoxolone methyl
  Other Names: RTA 402

SUMMARY:
This extended access study will assess the long-term safety and tolerability of bardoxolone methyl in qualified patients with pulmonary hypertension (PH) who previously participated in controlled clinical studies with bardoxolone methyl.

DETAILED DESCRIPTION:
This extended access study will assess the long-term safety and tolerability of bardoxolone methyl in qualified patients with pulmonary hypertension (PH) who previously participated in controlled clinical studies with bardoxolone methyl.

Qualified patients will receive 10 mg of bardoxolone methyl once daily until the drug is available through commercial channels or until patient withdrawal, whichever is sooner. Dose de-escalation (down to 5 mg) is permitted during the study, if indicated clinically.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-compliant patients who are participating in qualifying ongoing studies and have completed required End-of-Treatment and/or Follow-up visits in a prior clinical study with bardoxolone methyl

Exclusion Criteria:

* Participation in other investigational clinical studies involving interventional products being tested or used in a way different from the approved form or when used for an unapproved indication;
* Patients who have an ongoing SAE from a clinical study that is assessed by the investigator as related to bardoxolone methyl;
* Unwilling to practice acceptable methods of birth control (both males who have partners of childbearing potential and females of childbearing potential) while taking study drug;
* Women who are pregnant or breastfeeding;
* Patient is, in the opinion of the investigator, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason;
* Known hypersensitivity to any component of the study drug

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (96):
- United States (46):
  - Banner University Medical Center, Phoenix Advanced Lung Disease Institute, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - Cedars Sinai Medical Center, Beverly Hills, California
  - University of California San Diego, La Jolla, California
  - VA Healthcare System of Greater Los Angeles, Los Angeles, California
  - David Geffen School of Medicine UCLA, Los Angeles, California
  - University of California Davis Medical Center - Division of Pulmonary and Critical Care, Sacramento, California
  - Harbor - UCLA Medical Center, Torrance, California
  - University of Colorado Denver - Division of Pulmonary Sciences, Aurora, Colorado
  - Georgetown University Medical Center - Department of Rheumatology, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine, Miami, Florida
  - Cleveland Clinic of Florida, Weston, Florida
  - Augusta University, Augusta, Georgia
  - Piedmont-Georgia Lung, Austell, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Maine Medical Center - Division of Pulmonary and Critical Care Medicine, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - NYU Langone Medical Center, New York, New York
  - University of Rochester - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University of Cincinnati - Department of Internal Medicine Pulmonary, Critical Care & Sleep Medicine, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - The University of Texas - Health Science Center & Medical School at Houston, Houston, Texas
  - University of Texas Houston - Division of Rheumatology and Clinical Immunogenetics, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Aurora Health Care, Milwaukee, Wisconsin
- Argentina (6):
  - Centro Médico Dra de Salvo, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Instituto de Investigaciones Clínicas Mar Del Plata, Buenos Aires, Mar Del Plata
  - Instituto de Cardiologia de Corrientes Juana Francisca Cabral, Corrientes
  - Hospital Privado Centro Médico de Córdoba, Córdoba
  - Instituto Cardiovascular de Rosario, Rosario
  - Hospital Provincial Dr Jose Maria Cullen, Santa Fe
- Australia (4):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
- Belgium (2):
  - UZ Leuven, Leuven, Vlaams Brabant
  - Hospital Erasme, Brussels
- Brazil (3):
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Dia do Pulmão, Blumenau, Santa Catarina
  - Instituto do Coração - HCFMUSP, São Paulo
- Canada (4):
  - Peter Lougheed Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Centre Hospitalier de l'Université Laval, Sainte-Foy, Quebec
- Czechia (2):
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut klinicke a experimentalni mediciny, Prague
- Germany (3):
  - Universitatsklinkum Carl Gustav Carus an der Tu, Dresden
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Thorax Klinik, Heidelberg
- Israel (2):
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Japan (9):
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Kobe University Hospital, Kobe, Hyōgo
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Kyorin University Hospital, Tokyo, Mitaka-shi
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Chiba University Hospital, Chiba
  - Hokkaido University Hospital, Sapporo
  - Kurume University Medical Center, Sendai
  - National Cerebral and Cardiovascular Center, Suita
- Mexico (4):
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Instituto Nacional de Cardiologia Dr. Ignacio Chavez, Mexico City, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Nuevo León, Monterrey
  - Unidad de Investigación Clínica En Medicina SC, Monterrey, Nuevo León
- Vrije Universiteit Amsterdam, Amsterdam, North Holland, Netherlands
- Philippines (3):
  - Philippine Heart Center, Quezon City, National Capital Region
  - Makati Medical Center, Makati
  - Philippine General Hospital (PGH), Manila
- Spain (5):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Virgen de La Salud, Toledo
- United Kingdom (2):
  - Golden Jubilee National Hospital, Glasgow
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Bardoxolone Methyl: Participants who received bardoxolone methyl capsules (administered orally). Dosing started at 10 mg once daily (if enrolled under version 2.0, 2.1 [UK], 2.2 [Germany] of the protocol) or every other day (if enrolled under version 3.0, 3.1 [UK], 3.1 and 3.2 [Germany] of the protocol). For participants who began by dosing every other day, once daily dosing at 10 mg began at Week 4, unless contraindicated clinically. In Japan, participants began dosing at 5 mg once daily then dose-escalated to 10 mg at Week 4, unless contraindicated clinically.
Period: Overall Study
Arm/Group | Bardoxolone Methyl
Started | 261
Completed | 0
Not Completed | 261
Not completed — Adverse Event | 19
Not completed — Death | 14
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 26
Not completed — Administrative Reasons | 3
Not completed — Protocol specified withdrawal criterion | 1
Not completed — Study terminated by sponsor | 194

BASELINE CHARACTERISTICS:
Population: Safety population (all patients who received at least 1 dose of bardoxolone methyl)
Arm/Group | Bardoxolone Methyl
Number analyzed (Participants) | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61
  Not Hispanic or Latino | 200
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 204
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  Argentina | 23
  United States | 161
  Czechia | 3
  Japan | 12
  Philippines | 5
  United Kingdom | 3
  Spain | 8
  Canada | 6
  Netherlands | 2
  Belgium | 3
  Brazil | 4
  Mexico | 11
  Israel | 3
  Australia | 13
  Germany | 4

OUTCOME MEASURES:

1. Primary Outcome: Long Term Safety as Measured by Incidence and Severity of Adverse Events During the Duration of the Study
Description: Severity was defined using the following definitions: Mild: Symptoms causing no or minimal interference with usual social and functional activities; Moderate: Symptoms causing greater than minimal interference with usual social and functional activities; Severe: Symptoms causing inability to perform usual social and functional activities.
Time Frame: From time of first dose until the final visit, up to 172 weeks
Population: Safety population (all patients who received at least 1 dose of bardoxolone methyl)
Measure: Count of Participants; unit: Participants
Arm/Group | Bardoxolone Methyl
Number analyzed (Participants) | 261
Participants
  Number and percent of participants with at least one adverse event | 232
  Number and percent of participants with a related adverse event | 89
  Number and percent of participants with a serious adverse event | 106
  Number and percent of participants with worst adverse event severity of mild | 42
  Number and percent of participants with worst adverse event severity of moderate | 96
  Number and percent of participants with worst adverse event severity of severe | 94

ADVERSE EVENTS:
Time Frame: The time from the date of a participant's first dose to his or her last participation or event date, a maximum of 172 weeks
Description: All AEs and SAEs from the time of administration of the first dose until the final visit were to be reported. AEs and SAEs that occurred within 30 days after the last dose were considered treatment emergent. For SAEs, the investigator was to follow the patient until the SAE subsided or until the condition became chronic in nature, stabilized (in the case of persistent impairment), or the patient died.
Arm/Group | Bardoxolone Methyl
All-Cause Mortality (participants affected / at risk) | 17/261
Serious Adverse Events (participants affected / at risk) | 106/261
Other Adverse Events (participants affected / at risk) | 198/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bardoxolone Methyl (N=261)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (5)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (3)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Dilatation ventricular (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 7 (10)
Systolic dysfunction (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Dental cyst (Gastrointestinal disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Oesophageal motility disorder (Gastrointestinal disorders) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Complication associated with device (General disorders) | 1 (1)
Device related thrombosis (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2)
Oedema peripheral (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bursitis infective (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 4 (4)
Cellulitis staphylococcal (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1)
Ecthyma (Infections and infestations) | 1 (1)
Haemophilus infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2)
Infectious colitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Meningitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 13 (13)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 3 (4)
Septic shock (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Drug administration error (Injury, poisoning and procedural complications) | 1 (1)
Environmental exposure (Injury, poisoning and procedural complications) | 1 (1)
Eschar (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Norovirus test positive (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebellar artery thrombosis (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Lateral medullary syndrome (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Spinal epidural haematoma (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Vasculitis cerebral (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 13 (16)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haematoma (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bardoxolone Methyl (N=261)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 14
Palpitations (Cardiac disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 41
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 31
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 6
Fatigue (General disorders) | 19
Non-cardiac chest pain (General disorders) | 10
Oedema peripheral (General disorders) | 16
Pyrexia (General disorders) | 8
Bronchitis (Infections and infestations) | 21
Cellulitis (Infections and infestations) | 8
Conjunctivitis (Infections and infestations) | 10
Herpes zoster (Infections and infestations) | 9
Influenza (Infections and infestations) | 14
Lower respiratory tract infection (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 13
Pneumonia (Infections and infestations) | 11
Respiratory tract infection (Infections and infestations) | 9
Sinusitis (Infections and infestations) | 22
Upper respiratory tract infection (Infections and infestations) | 51
Urinary tract infection (Infections and infestations) | 30
Arthropod bite (Injury, poisoning and procedural complications) | 6
Brain natriuretic peptide increased (Investigations) | 6
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 21
Weight decreased (Investigations) | 16
Decreased appetite (Metabolism and nutrition disorders) | 15
Hypokalaemia (Metabolism and nutrition disorders) | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 7
Vitamin D deficiency (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 33
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17
Pain in jaw (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 22
Headache (Nervous system disorders) | 26
Syncope (Nervous system disorders) | 9
Insomnia (Psychiatric disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 9
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 7
Skin ulcer (Skin and subcutaneous tissue disorders) | 7
Hypotension (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (5):
  • Study Protocol: US Protocol (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT03068130/Prot_000.pdf
  • Study Protocol: Japan Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT03068130/Prot_001.pdf
  • Study Protocol: UK Protocol (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT03068130/Prot_002.pdf
  • Study Protocol: Germany Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT03068130/Prot_003.pdf
  • Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03068130/SAP_004.pdf